CLINICAL TRIAL: NCT00774020
Title: A 6 Months, Open-Label Phase IV Study to Confirm the Safety and Efficacy of Single Intravenous Dose of 5 mg Zoledronic Acid for the Patients of Paget's Disease of Bone (PDB) in China
Brief Title: Efficacy and Safety of Single Dose of 5 mg Zoledronic Acid in Chinese Patients With Paget's Disease of Bone (PDB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446K2419
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Paget's Disease of Bone
Keywords: Paget's Disease of Bone; Serum Alkaline Phosphatase
MeSH Terms: conditions — Osteitis Deformans | interventions — Zoledronic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — 5mg, i.v. single dose

SUMMARY:
The purpose of this study is to document the efficacy and safety profiles of single intravenous dose of 5 mg zoledronic acid for the Chinese patients of Paget's Disease of Bone (PDB).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PDB by radiological reports
* Serum Alkaline Phosphatase level (SAP) at least two times the upper limit of the normal (ULN)

Exclusion Criteria:

* History of hypersensitivity to the active substance or to any of the excipients or to any bisphosphonates;
* History of malignancy of any organ system
* Severe liver or bladder disease;
* Calculated creatinine clearance < 35 mL/min at baseline;
* Hypocalcaemia;
* Patients with pre-existing dental diseases or who predict to have dental surgeries during the study;
* Evidence of vitamin D deficiency.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10-30 (Actual); Primary Completion 2011-01-14 (Actual); Study Completion 2011-01-14 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieve therapeutic response (a reduction of at least 75% from baseline in total Serum Alkaline Phosphatase (SAP) excess or normalization of SAP. | at the end of 3 months and 6 months

SECONDARY OUTCOMES:
The percent change from baseline in total Serum Alkaline Phosphatase (SAP). | at the end of 3 months and 6 months
The percent change from baseline in serum cross-linked C-telopeptide of type I collagen (CTX). | at the end of 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative site, Guangzhou
  - Novartis Investigative site, Nanjing
  - Novartis Investigative site, Shanghai